CLINICAL TRIAL: NCT02222610
Title: A Randomized, Active-Controlled, Phase II Study of the Efficacy and Tolerability of Intravitreal Injections of Ranibizumab Compared to Intravitreal Injections of Ranibizumab Combined With Targeted Retinal Photocoagulation in Subjects With Radiation Retinopathy (RRR Study).
Brief Title: Study of the Efficacy and Tolerability of Intravitreal Injections of Ranibizumab Compared to Intravitreal Injections of Ranibizumab Combined With Targeted Retinal Photocoagulation to Treat Radiation Retinopathy.
Acronym: RRR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Greater Houston Retina Research (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML29236
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Radiation Retinopathy
Keywords: Radiation Retinopathy
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Experimental): Subject's will receive monthly treatment of an intravitreal injection of 0.5 mg ranibizumab for 48 weeks.
  Starting at week 52, subject's will enter a treat & extend regime, if a subject achieves a "dry" macula. For a macula to be considered "dry" persistent or recurrent fluid must be resolved on spectral domain (SD)-optical coherence tomography (OCT). The interval between injections will not exceed 12 weeks. After a subject is extended beyond 4-weeks & develops recurrent disease activity, the eye is treated & the treatment interval for the next visit is reduced by 1 week, compared to the previous treatment interval. The interval between treatments will be reduced by 1-week intervals until a dry macula is again established. Once a dry macula is again achieved, the interval between visits will be extended by 1-week intervals again.
  Interventions: Drug: 0.5 mg ranibizumab
- Cohort B (Experimental): Subject's receive monthly treatment of IVT of 0.5 mg ranibizumab for 48 weeks. 1 week after the initial dose of IVT ranibizumab, the subject will have peripheral targeted-retinal photocoagulation (TRP) to areas of peripheral retinal ischemia based on 120° or greater wide field angiography. After the first session of TRP, subjects will have a repeat wide field angiogram at 12 weeks & 24 weeks & will receive additional TRP as needed (PRN) to areas of peripheral retinal ischemia.
  Starting at week 52, subject's will enter a treat & extend regime as described in cohort A.
  Interventions: Drug: 0.5 mg ranibizumab; Procedure: Targeted Retinal Photocoagulation (TRP)
- Cohort C (Experimental): Subject's will receive 3 consecutive monthly doses of IVT 0.5 mg ranibizumab followed by PRN treatment with 0.5 mg ranibizumab intravitreal injection. 1 week after the initial dose of IVT ranibizumab, the subject will have peripheral targeted-retinal photocoagulation (TRP) to areas of peripheral retinal ischemia. After the first session of TRP, subjects will have a repeat wide field angiogram at 12 weeks & 24 weeks & will receive additional TRP as needed (PRN) to areas of peripheral retinal ischemia.
  Starting at week 52, subject's will enter a treat & extend regime as described in cohort A.
  Interventions: Drug: 0.5 mg ranibizumab; Procedure: Targeted Retinal Photocoagulation (TRP)

INTERVENTIONS:
Drug: 0.5 mg ranibizumab
  Other Names: Lucentis
Procedure: Targeted Retinal Photocoagulation (TRP) — TRP to areas of retinal ischemia
  Arms: Cohort B; Cohort C

SUMMARY:
The purpose of this study is to assess the tolerability and efficacy of ranibizumab treatment administered in subjects with radiation retinopathy

DETAILED DESCRIPTION:
RRR is a phase II, randomized, multicenter, clinical study to assess the tolerability and efficacy of ranibizumab treatment administered in subjects with radiation retinopathy. Subjects will be randomized into one of 3 arms; intravitreal (IVT) monthly vs. ranibizumab treatment administered IVT monthly combined with peripheral targeted photocoagulation vs. ranibizumab treatment administered IVT for three months followed by as needed treatment of ranibizumab combined with peripheral targeted photocoagulation over 48 weeks. From week 52 to week 101, all 3 treatment arms will employ a treat and extend protocol for IVT ranibizumab treatment.

ELIGIBILITY:
Inclusion Criteria

Subjects will be eligible to participate if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Active radiation retinopathy resulting from any form of radiation treatment performed within the last 3 years. Radiation retinopathy is defined as any of the following: retinal hemorrhages, exudates, edema, and/or neovascularization, not attributable to other causes.
* Best Corrected Visual Acuity (BCVA) of 20/25-20/400 in the study eye

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

* Pregnancy (verified by positive pregnancy test) or lactation
* Premenopausal women not using adequate methods of contraception. The following are considered effective means of contraception: surgical sterilization, use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an intrauterine device (IUD), or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Participation in any other simultaneous medical investigation or trial
* Previous participation in any studies involving investigational drugs within 30 days before Day 0 (excluding vitamins and minerals).
* History of allergy fluorescein, not amenable to treatment
* Previous intravitreal treatment with any anti-vascular endothelial growth factor (VEGF) drug within 60 days of Day 0
* Previous intravitreal or subconjunctival treatment with cortical steroids within 90 days of Day 0
* History of vitrectomy
* History of treatment with more than one form of radiation to the eye (e.g. proton beam therapy and plaque therapy).
* Subjects who have more than 7 disc diameters of ischemia in the central macula that would hinder visual acuity improvement
* History of panretinal photocoagulation treatment in the study eye.
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed
* Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could:

  * Require medical or surgical intervention during the 12 month study period to prevent or treat visual loss that might result from that condition.
  * Contribute to loss of at least 2 Snellen equivalent lines of BCVA over the 12-month study period, if allowed to progress untreated.
* Active intraocular inflammation (grade 2+ or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (stage 3 or 4) in the study eye.
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.
* Aphakia or absence of the posterior capsule in the study eye.
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding Day 0.
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure (IOP) > 30 mmHg despite treatment with anti-glaucoma medication).
* History of glaucoma-filtering surgery in the study eye
* History of corneal transplant in the study eye
* Uncontrolled blood pressure (defined as systolic and/or diastolic > 180/110 mmHg while subject is seated). If the subject's initial reading exceeds these values, a second reading may be taken at least 30 minutes later. If the subject requires antihypertensive medication, the subject can become eligible if medication is taken continuously for at least 14 days prior to Day 0 and blood pressure is less that 180/110 mmHg.
* New diagnosis of atrial fibrillation not managed by subject's primary care physician or cardiologist within 3 months of Day 0.
* History of stroke within the last 3 months of Day 0.
* History of myocardial infarction within 3 months of Day 0.
* History of other disease, metabolic dysfunction, or physical examination finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or renders the subject at high risk for treatment complications.
* Current treatment for active systemic infection
* Active malignancy other than uveal melanoma
* Presence of metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Schefler, MD, Principal Investigator — Retina Consultants Houston
Locations (4):
- United States (4):
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston/The Medical Center, Houston, Texas
  - Retina Consultants of Houston, Katy, Texas
  - Retina Consultants of Houston, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jampol LM, Moy CS, Murray TG, Reynolds SM, Albert DM, Schachat AP, Diddie KR, Engstrom RE Jr, Finger PT, Hovland KR, Joffe L, Olsen KR, Wells CG; Collaborative Ocular Melanoma Study Group (COMS Group). The COMS randomized trial of iodine 125 brachytherapy for choroidal melanoma: IV. Local treatment failure and enucleation in the first 5 years after brachytherapy. COMS report no. 19. Ophthalmology. 2002 Dec;109(12):2197-206. doi: 10.1016/s0161-6420(02)01277-0. PMID 12466159
- [Background] Melia BM, Abramson DH, Albert DM, Boldt HC, Earle JD, Hanson WF, Montague P, Moy CS, Schachat AP, Simpson ER, Straatsma BR, Vine AK, Weingeist TA; Collaborative Ocular Melanoma Study Group. Collaborative ocular melanoma study (COMS) randomized trial of I-125 brachytherapy for medium choroidal melanoma. I. Visual acuity after 3 years COMS report no. 16. Ophthalmology. 2001 Feb;108(2):348-66. doi: 10.1016/s0161-6420(00)00526-1. PMID 11158813
- [Background] Gunduz K, Shields CL, Shields JA, Cater J, Freire JE, Brady LW. Radiation retinopathy following plaque radiotherapy for posterior uveal melanoma. Arch Ophthalmol. 1999 May;117(5):609-14. doi: 10.1001/archopht.117.5.609. PMID 10326957
- [Background] Finger PT, Chin KJ. High-dose (2.0 mg) intravitreal ranibizumab for recalcitrant radiation retinopathy. Eur J Ophthalmol. 2013 Nov-Dec;23(6):850-6. doi: 10.5301/ejo.5000333. Epub 2013 Jun 28. PMID 23813109
- [Background] Finger PT, Chin KJ. Intravitreous ranibizumab (lucentis) for radiation maculopathy. Arch Ophthalmol. 2010 Feb;128(2):249-52. doi: 10.1001/archophthalmol.2009.376. No abstract available. PMID 20142553
- [Background] Finger PT, Chin KJ. Antivascular endothelial growth factor bevacizumab for radiation optic neuropathy: secondary to plaque radiotherapy. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):789-98. doi: 10.1016/j.ijrobp.2010.11.075. Epub 2011 Jan 27. PMID 21277107
- [Background] Finger PT, Mukkamala SK. Intravitreal anti-VEGF bevacizumab (Avastin) for external beam related radiation retinopathy. Eur J Ophthalmol. 2011 Jul-Aug;21(4):446-51. doi: 10.5301/EJO.2011.6213. PMID 21218391
- [Background] Mason JO 3rd, Albert MA Jr, Persaud TO, Vail RS. Intravitreal bevacizumab treatment for radiation macular edema after plaque radiotherapy for choroidal melanoma. Retina. 2007 Sep;27(7):903-7. doi: 10.1097/IAE.0b013e31806e6042. PMID 17891015
- [Background] Finger PT. Radiation retinopathy is treatable with anti-vascular endothelial growth factor bevacizumab (Avastin). Int J Radiat Oncol Biol Phys. 2008 Mar 15;70(4):974-7. doi: 10.1016/j.ijrobp.2007.11.045. PMID 18313522
- [Background] Finger PT, Chin K. Anti-vascular endothelial growth factor bevacizumab (avastin) for radiation retinopathy. Arch Ophthalmol. 2007 Jun;125(6):751-6. doi: 10.1001/archopht.125.6.751. PMID 17562985
- [Background] Gupta A, Muecke JS. Treatment of radiation maculopathy with intravitreal injection of bevacizumab (Avastin). Retina. 2008 Jul-Aug;28(7):964-8. doi: 10.1097/IAE.0b013e3181706302. PMID 18698298
- [Background] Shields CL, Demirci H, Dai V, Marr BP, Mashayekhi A, Materin MA, Manquez ME, Shields JA. Intravitreal triamcinolone acetonide for radiation maculopathy after plaque radiotherapy for choroidal melanoma. Retina. 2005 Oct-Nov;25(7):868-74. doi: 10.1097/00006982-200510000-00009. PMID 16205566
- [Background] Finger PT, Kurli M. Laser photocoagulation for radiation retinopathy after ophthalmic plaque radiation therapy. Br J Ophthalmol. 2005 Jun;89(6):730-8. doi: 10.1136/bjo.2004.052159. PMID 15923510
- [Background] Kinyoun JL. Long-term visual acuity results of treated and untreated radiation retinopathy (an AOS thesis). Trans Am Ophthalmol Soc. 2008;106:325-35. PMID 19277244
- [Background] Hykin PG, Shields CL, Shields JA, Arevalo JF. The efficacy of focal laser therapy in radiation-induced macular edema. Ophthalmology. 1998 Aug;105(8):1425-9. doi: 10.1016/S0161-6420(98)98023-X. PMID 9709753
- [Background] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Regillo CD, Brown DM, Abraham P, Yue H, Ianchulev T, Schneider S, Shams N. Randomized, double-masked, sham-controlled trial of ranibizumab for neovascular age-related macular degeneration: PIER Study year 1. Am J Ophthalmol. 2008 Feb;145(2):239-248. doi: 10.1016/j.ajo.2007.10.004. PMID 18222192
- [Background] Brown DM, Michels M, Kaiser PK, Heier JS, Sy JP, Ianchulev T; ANCHOR Study Group. Ranibizumab versus verteporfin photodynamic therapy for neovascular age-related macular degeneration: Two-year results of the ANCHOR study. Ophthalmology. 2009 Jan;116(1):57-65.e5. doi: 10.1016/j.ophtha.2008.10.018. PMID 19118696
- [Background] Boyer DS, Heier JS, Brown DM, Francom SF, Ianchulev T, Rubio RG. A Phase IIIb study to evaluate the safety of ranibizumab in subjects with neovascular age-related macular degeneration. Ophthalmology. 2009 Sep;116(9):1731-9. doi: 10.1016/j.ophtha.2009.05.024. Epub 2009 Jul 29. PMID 19643495
- [Derived] Yu HJ, Fuller D, Anand R, Fuller T, Munoz J, Moore C, Kim RS, Schefler AC; RRR Study Group. Two-year results for ranibizumab for radiation retinopathy (RRR): a randomized, prospective trial. Graefes Arch Clin Exp Ophthalmol. 2022 Jan;260(1):47-54. doi: 10.1007/s00417-021-05281-2. Epub 2021 Aug 31. PMID 34463842

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Cohort A: Subject's will receive monthly treatment of an intravitreal injection of 0.5 mg ranibizumab for 48 weeks.
  Starting at week 52, subject's will enter a treat & extend regime, if a subject achieves a "dry" macula. For a macula to be considered "dry" persistent or recurrent fluid must be resolved on SD-OCT. The interval between injections will not exceed 12 weeks. After a subject is extended beyond 4-weeks & develops recurrent disease activity, the eye is treated & the treatment interval for the next visit is reduced by 1 week, compared to the previous treatment interval. The interval between treatments will be reduced by 1-week intervals until a dry macula is again established. Once a dry macula is again achieved, the interval between visits will be extended by 1-week intervals again.
  0.5 mg ranibizumab
- Cohort B: Subject's receive monthly treatment of intravitreal (IVT) 0.5 mg ranibizumab for 48 weeks. 1 week after the initial dose of IVT ranibizumab, the subject will have peripheral targeted-retinal photocoagulation (TRP) to areas of peripheral retinal ischemia based on 120° or greater wide field angiography. After the first session of TRP, subjects will have a repeat wide field angiogram at 12 weeks & 24 weeks & will receive additional TRP as needed (PRN) to areas of peripheral retinal ischemia.
  Starting at week 52, subject's will enter a treat & extend regime as described in cohort A.
  0.5 mg ranibizumab
  Targeted Retinal Photocoagulation (TRP): TRP to areas of retinal ischemia
- Cohort C: Subject's will receive 3 consecutive monthly doses of IVT 0.5 mg ranibizumab followed by PRN treatment with 0.5 mg ranibizumab intravitreal injection. 1 week after the initial dose of IVT ranibizumab, the subject will have peripheral targeted-retinal photocoagulation (TRP) to areas of peripheral retinal ischemia. After the first session of TRP, subjects will have a repeat wide field angiogram at 12 weeks & 24 weeks & will receive additional TRP as needed (PRN) to areas of peripheral retinal ischemia.
  Starting at week 52, subject's will enter a treat & extend regime as described in cohort A.
  0.5 mg ranibizumab
  Targeted Retinal Photocoagulation (TRP): TRP to areas of retinal ischemia
Period: Baseline to W48
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 8; 8 eyes | 16; 16 eyes | 16; 16 eyes
Completed | 8; 8 eyes | 14; 14 eyes | 15; 15 eyes
Not Completed | 0; 0 eyes | 2; 2 eyes | 1; 1 eyes
Period: Baseline to W104
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 8; 8 eyes | 16; 16 eyes | 16; 16 eyes
Completed | 8; 8 eyes | 11; 11 eyes | 10; 10 eyes
Not Completed | 0; 0 eyes | 5; 5 eyes | 6; 6 eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Cohort B: Subject's receive monthly treatment of IVT of 0.5 mg ranibizumab for 48 weeks. 1 week after the initial dose of IVT ranibizumab, the subject will have peripheral targeted-retinal photocoagulation (TRP) to areas of peripheral retinal ischemia based on 120° or greater wide field angiography. After the first session of TRP, subjects will have a repeat wide field angiogram at 12 weeks & 24 weeks & will receive additional TRP as needed (PRN) to areas of peripheral retinal ischemia.
  Starting at week 52, subject's will enter a treat & extend regime as described in cohort A.
  0.5 mg ranibizumab
  Targeted Retinal Photocoagulation (TRP): TRP to areas of retinal ischemia
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 8 | 16 | 16 | 40
Number analyzed (Eyes) | 8 | 16 | 16 | 40
Age, Continuous [Mean (Full Range); unit: years] | 66.125 [52 to 76] | 54.813 [29 to 72] | 60.438 [21 to 81] | 57 [22 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 16
  Male | 3 | 10 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 16 | 15 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 15 | 16 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 16 | 16 | 40
Best-Corrected Visual Acuity [Mean (Full Range); unit: letters] — Early Treatment Diabetic Retinopathy Study (ETDRS) Best-Corrected Visual Acuity (BCVA) utilizes the ETDRS visual acuity chart to measure vision in clinical trials. Standard unit of measure is the number of letters subjects are able to read on the chart.
  letters | 60.875 [36 to 81] | 55.813 [27 to 76] | 55.375 [23 to 74] | 56.7 [23 to 81]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity at 104 Weeks From Day 0.
Description: Early Treatment Diabetic Retinopathy Study (ETDRS) Best-Corrected Visual Acuity (BCVA) utilizes the ETDRS visual acuity chart to measure vision in clinical trials. Standard unit of measure is the number of letters subjects are able to read on the chart.
Time Frame: 104 weeks
Population: Subjects analyzed only include those that completed the W104 visit.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 8 | 11 | 10
letters | -1.9 (7.4) | -3.9 (16.5) | 1.3 (11.8)

2. Secondary Outcome: The Mean Number of Intravitreal Injections Required Per Subject Per Cohort.
Time Frame: 104 weeks
Measure: Mean (Full Range); unit: injections
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 8 | 16 | 16
injections | 22.2 [19 to 25] | 18.5 [11 to 25] | 16.1 [6 to 26]

3. Secondary Outcome: Percentage of Subjects With Retinal Hemorrhage at 104 Weeks.
Time Frame: 104 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 8 | 16 | 16
Participants | 1 | 0 | 3

4. Secondary Outcome: Percentage of Subjects With Intraretinal Exudates on Fundus Examination at Week 104.
Time Frame: 104 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 8 | 16 | 16
Participants | 1 | 2 | 5

5. Secondary Outcome: Mean Change in Central Mean Thickness According to Spectral-domain Optical Coherence Tomography at Week 104 Compared to Baseline.
Description: Spectral-domain optical coherence tomography (SD-OCT) is a common imaging modality used to visualize the layers of the macula. Central mean thickness (CMT) is the length in microns from the internal limiting membrane to Bruch's membrane.
Time Frame: 104 weeks
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 8 | 16 | 16
micrometers | -8.5 (216.7) | -87 (174.8) | -74.6 (176.7)

ADVERSE EVENTS:
Time Frame: Baseline through 104 weeks
Arm/Group | Cohort A | Cohort B | Cohort C
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/16 | 1/16
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/16 | 5/16
Other Adverse Events (participants affected / at risk) | 3/8 | 7/16 | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=8) | Cohort B (N=16) | Cohort C (N=16)
Acute Chronic Diastolic Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Chronic Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Broken Wrist (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Central Retinal Artery Occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Recurrence of Choroidal Melanoma (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Metastatic Uveal Melanom (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Pancreatitis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Worsening of Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=8) | Cohort B (N=16) | Cohort C (N=16)
Corneal Abrasion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Increased Cup-to-Disc Rratio (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Ocular Irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Posterior Capsular Opacification (Eye disorders) | 0 (0) | 1 (1) | 2 (3)
Posterior Vitreous Detachment (Eye disorders) | 1 (1) | 3 (3) | 1 (1)
Subconjunctival Hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Worsening of Cataracts (Eye disorders) | 2 (2) | 5 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-07-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02222610/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT02222610/SAP_001.pdf